CLINICAL TRIAL: NCT06741592
Title: The Effect of Different Irrigation Activation Methods Preferred During Root Canal Treatment On Postoperative Pain: A Randomized Clinical Trial
Brief Title: Postoperative Pain in Endodontic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Seca MUTLU, Research Assistant, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ODU-MUTLU-001
Record Dates: First submitted 2024-12-12; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Endodontic Disease; Postoperative Pain
Keywords: EDDY; Irrigation Activation; Passive Ultrasonic Irrigation
MeSH Terms: conditions — Dental Pulp Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EDDY Group (Experimental): The effect of the EDDY device, preferred for root canal irrigation activation, on postoperative pain formation
  Interventions: Device: EDDY Group
- PUI Group (Experimental): The effect of the passive ultrasonic activation method, preferred for root canal irrigation activation, on postoperative pain formation
  Interventions: Device: PUI Group
- Control Group (No Intervention): Root canal treatment performed with conventional irrigation without the use of any activation method

INTERVENTIONS:
Device: EDDY Group — The EDDY activation of the irrigation solutions used is performed to achieve root canal disinfection and enhance antibacterial effectiveness once the root canal preparation is completed.
  Arms: EDDY Group
Device: PUI Group — The passive ultrasonic activation of the irrigation solutions used is performed to achieve root canal disinfection and enhance antibacterial effectiveness once the root canal preparation is completed.
  Arms: PUI Group

SUMMARY:
The goal of this clinical trial is to evaluate the change in postoperative pain in mandibular premolar and first molar teeth with asymptomatic apical periodontitis when using EDDY and passive ultrasonic irrigation activation methods.

The null hypothesis is: "There is no difference in postoperative pain after root canal treatment between the irrigation activation systems in mandibular first molars and premolar teeth."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 55 years, medically healthy, and free from systemic diseases.
* Patients without pregnancy or breastfeeding status.
* Patients diagnosed with asymptomatic apical periodontitis confirmed through radiographic and clinical examination.
* Patients not having a regular intake of analgesic or anti-inflammatory drugs within the last 12 hours.
* Patients lacking a history of drug allergies.
* Teeth free from calcifications, resorptions, periodontal problems, incomplete root development, a history of endodontic treatment, traumatic occlusion, or severe coronal destruction.
* Teeth with a root canal curvature of 5° or less.
* Mandibular premolars and first molars.

Exclusion Criteria:

* Teeth where the apical area could not be reached with a #8K file.
* Teeth with an apical diameter larger than #20K file.
* Patients with a Periapical Index (PAI) score of 1 or 2.
* Teeth having extra canals.
* Teeth requiring a second local anesthesia during treatment.
* Teeth where a file fractured within the canal during preparation.
* Vital teeth.
* Patients reporting preoperative pain.
* Teeth showing clinical symptoms such as percussion or palpation sensitivity.
* Teeth with persistent purulent discharge.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 8th hour
  Prior to treatment, patients were instructed in detail on how to complete the VAS (Visual Analog Scale). Patients were asked to mark their pain levels on a 10 cm line based on the severity of pain experienced after the procedure. Pain intensity was numerically documented on a scale of 0 to 10. 0 is described as no pain number, 10 is described as the highest pain number.
Postoperative Pain | 12th hour
  Prior to treatment, patients were instructed in detail on how to complete the VAS (Visual Analog Scale). Patients were asked to mark their pain levels on a 10 cm line based on the severity of pain experienced after the procedure. Pain intensity was numerically documented on a scale of 0 to 10. 0 is described as no pain number, 10 is described as the highest pain number.
Postoperative Pain | 24th hour
  Prior to treatment, patients were instructed in detail on how to complete the VAS (Visual Analog Scale). Patients were asked to mark their pain levels on a 10 cm line based on the severity of pain experienced after the procedure. Pain intensity was numerically documented on a scale of 0 to 10. 0 is described as no pain number, 10 is described as the highest pain number.
Postoperative Pain | 48th hour
  Prior to treatment, patients were instructed in detail on how to complete the VAS (Visual Analog Scale). Patients were asked to mark their pain levels on a 10 cm line based on the severity of pain experienced after the procedure. Pain intensity was numerically documented on a scale of 0 to 10. 0 is described as no pain number, 10 is described as the highest pain number.
Postoperative Pain | 7th day
  Prior to treatment, patients were instructed in detail on how to complete the VAS (Visual Analog Scale). Patients were asked to mark their pain levels on a 10 cm line based on the severity of pain experienced after the procedure. Pain intensity was numerically documented on a scale of 0 to 10. 0 is described as no pain number, 10 is described as the highest pain number.

CONTACTS AND LOCATIONS:
Overall Officials: Seca MUTLU, Principal Investigator — Ordu University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Ordu University, Ordu, Karadeniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No